CLINICAL TRIAL: NCT07169864
Title: An Exploratory Self-Controlled Study on the Preventive Effect of the Simple Surgical Glove Compression Technique Against Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Simple Surgical Glove Compression to Prevent Chemotherapy-Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinsong Lu (Other)
Responsible Party: Sponsor-Investigator, Jinsong Lu, Chief of Department of Breast Surgery, RenJi Hospital
Organization: RenJi Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LY2025-246-C
Record Dates: First submitted 2025-08-27; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Chemotherapy Induced Peripheral Neuropathy (CIPN); Neoadjuvant Therapy
Keywords: Utidelone; CIPN; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group with surgical glove compression applied to the dominant hand (Experimental)
  Interventions: Procedure: Simple Surgical Glove Compression Technique

INTERVENTIONS:
Procedure: Simple Surgical Glove Compression Technique — Patients will wear surgical gloves of smaller size than the patient's hand, on the dominant hand from 15 minutes before the start of each neoadjuvant chemotherapy infusion until 15 minutes after the end of infusion (total of 90 minutes). The non-dominant hand will serve as the untreated control.

SUMMARY:
To evaluate the preventive efficacy of a simple surgical glove compression technique in reducing the incidence and severity of Chemotherapy Induced Peripheral Neuropathy among patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Histologically confirmed primary invasive breast cancer;
* Planned to receive ≥ 8 weeks of weekly neoadjuvant chemotherapy (utidelone plus cisplatin);
* ECOG performance status: 0-1;

Exclusion Criteria:

* Distant metastasis;
* Presence of sensory or motor neurological disorders, or symptoms related to peripheral neuropathy with CTCAE grade ≥ 2, or currently receiving medication for peripheral neuropathy;
* Conditions affecting limb function;
* Known allergy to glove materials (e.g., latex)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the functional assessment of cancer therapy/gynaecologic oncology group-neurotoxicity (FACT/GOG-Ntx) subscale score(range:-44to44; higher scores indicate better neurotoxicity-related quality of life). | From baseline (prior to neoadjuvant chemotherapy) to after 8 weeks of neoadjuvant chemotherapy in breast cancer

SECONDARY OUTCOMES:
Change in scores and the sum score of four hand-related items of the FACT/GOG-Ntx subscale (range: -16to+16; higher scores indicate better neurotoxicity-related quality of life). | From baseline (prior to neoadjuvant chemotherapy) to after 8 weeks of neoadjuvant chemotherapy in breast cancer
The overall change in the FACT/GOG-Ntx subscale score (range: -44to44; higher scores indicate better neurotoxicity-related quality of life) | From baseline to the end of neoadjuvant chemotherapy and 6 months after completion of neoadjuvant chemotherapy
Incidence of CIPN as determined by changes in tactile sensitivity assessed with the Semmes-Weinstein monofilament test | From baseline to the end of and 6 months after completion of neoadjuvant chemotherapy
Incidence of CIPN according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | From baseline to the end of and 6 months after completion of neoadjuvant chemotherapy
Changes in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) scores (range: -12to12, higher scores on functional and global health domains indicate better quality of life,; -84to84; while higher | At baseline (prior to initiation of neoadjuvant chemotherapy), at 8 weeks of neoadjuvant chemotherapy, at 2 weeks after completion of neoadjuvant chemotherapy, and at 6 months after completion of neoadjuvant chemotherapy.
Changes in the maximum width and height of the lunula of each finger | At baseline (prior to initiation of neoadjuvant chemotherapy), at 8 weeks of neoadjuvant chemotherapy, at 2 weeks after completion of neoadjuvant chemotherapy, and at 6 months after completion of neoadjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China